CLINICAL TRIAL: NCT00266513
Title: Studies of Disorders in Antibody Production and Related Primary Immunodeficiency States
Status: Terminated | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 060049; 06-I-0049
Record Dates: First submitted 2005-12-16; First posted 2005-12-16 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2013-07-11

CONDITIONS: Hyper-IgM Syndrome; Ectodermal Dysplasia
Keywords: CD40 Ligand; Nemo; Genetics; Hyper-IGM; Ectodermal Dysplasia; CVID; Hyper-IgM Syndrome; Primary Immune Deficiency Disorders; Common Variable Immune Deficiency
MeSH Terms: conditions — Hyper-IgM Immunodeficiency Syndrome; Ectodermal Dysplasia; Incontinentia Pigmenti; Primary Immunodeficiency Diseases; Common Variable Immunodeficiency

SUMMARY:
This study investigates gene abnormalities in Primary Immune Deficiency(PID) with a goal of improving the diagnosis and treatment of patients.

The specific disorders include:

1. X linked hyper IgM Syndrome which is caused by an abnormality in the CD40L gene.
2. NEMO associated immune deficiency which is caused by an abnormality in a gene called NEMO.
3. Common variable immunodeficiency (CVID) which has an unknown genetic basis.
4. Other disorders of immunoglobulin production.

This study will:

1. Better characterize the clinical features of CD40 L deficiency and NEMO associated immune deficiency and other related primary immune deficiency syndromes.
2. Determine the frequency of CD40 L and Nemo abnormalities.
3. Determine whether particular abnormalities in these genes are associated with more of less severe illness or with specific symptoms.
4. Explore the basic mechanism by which these altered genes cause immune dysfunction.
5. Identify other genes causing low immune globulin levels and related primary immune deficient states.

DETAILED DESCRIPTION:
This protocol is designed to study the genetics and pathophysiology of Hyper-IgM syndrome, NEMO associated immune deficiency, patients with related primary immune deficiency disorders, and the blood relatives of immunodeficient patients. Patients will undergo evaluations that include history/physical, blood sampling, genetic testing, and possible tissue sampling. Among the aims of this protocol are to better understand genetic factors that lead to defects in host defense, and to use modern and evolving methods in molecular and cellular biology to elucidate the pathogenesis of these diseases. A better understanding of primary immunodeficiency could allow for the rational development of novel therapies for such diseases and to benefit future patients, but it might not benefit current patients directly. Routine follow-up may occur every six months - with evaluation and blood sampling. Under some circumstances, we may provide treatment that relates to the immune deficiency. These treatments will follow standard medical practice.

ELIGIBILITY:
* INCLUSION CRITERIA:

All patients must have a known or suspected immune defect with hyper-IgM syndrome and/or disorders of immunoglobulin production. There will be no limit on age, sex, race, or disability. Normal volunteers must be healthy adults between the age of 18 and 70 years. All study participants enrolled on to this study must agree to allow PI to store research samples. Refusal to let PI store samples may lead to withdrawal fro this specific study.

EXCLUSION CRITERIA:

The presence of an acquired abnormality, which leads to immune defects, such as HIV, chemotherapy, and malignancy are general exclusion criteria. Refusal to let us store samples may lead to withdrawal from this specific study. Other factors, which are in the judgment of the Principal Investigator PI that may interfere with patient evaluation or determine to pose an added risk for study participants are also criteria for exclusion.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2005-12-14; Study Completion 2013-07-11

CONTACTS AND LOCATIONS:
Overall Officials: Ashish K Jain, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Durandy A, Revy P, Imai K, Fischer A. Hyper-immunoglobulin M syndromes caused by intrinsic B-lymphocyte defects. Immunol Rev. 2005 Feb;203:67-79. doi: 10.1111/j.0105-2896.2005.00222.x. PMID 15661022
- [Background] Jain A, Atkinson TP, Lipsky PE, Slater JE, Nelson DL, Strober W. Defects of T-cell effector function and post-thymic maturation in X-linked hyper-IgM syndrome. J Clin Invest. 1999 Apr;103(8):1151-8. doi: 10.1172/JCI5891. PMID 10207167
- [Background] Durandy A, Revy P, Fischer A. Human models of inherited immunoglobulin class switch recombination and somatic hypermutation defects (hyper-IgM syndromes). Adv Immunol. 2004;82:295-330. doi: 10.1016/S0065-2776(04)82007-8. No abstract available. PMID 14975260